CLINICAL TRIAL: NCT01229735
Title: A Randomized, Open-label, Parallel Group, Multi-center, Comparative, Phase IV Trial of Levetiracetam (LEV) Versus Topiramate (TPM) as Adjunctive Therapy to Evaluate Efficacy and Safety in Subjects With Refractory Partial Onset Seizures
Brief Title: Levetiracetam Versus Topiramate as Adjunctive Therapy to Evaluate Efficacy and Safety in Subjects With Refractory Partial Onset Seizures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Korea Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N01353
Record Dates: First submitted 2010-10-26; First posted 2010-10-28 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-07

CONDITIONS: Epilepsy
Keywords: levetiracetam; topiramate; epilepsy; partial seizures
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Levetiracetam; Topiramate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levetiracetam (Experimental): 250 mg and 500 mg levetiracetam tablet; titration from 1000 mg/day (500 mg bid) to 3000 mg/day (1500 mg bid) levetiracetam with treatment duration up to 52 weeks
  Interventions: Drug: Levetiracetam
- Topiramate (Active Comparator): 25 mg and 100 mg topiramate tablet; titration from 100 mg/day (50 mg bid) to 400 mg/day (200 mg bid) topiramate with treatment duration up to 52 weeks
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Levetiracetam — 250 mg and 500 mg levetiracetam tablet 1000 mg/day (500 mg bid) levetiracetam (maximum to 3000 mg/day) Duration: maximum 52 weeks
  Other Names: Keppra
  Arms: Levetiracetam
Drug: Topiramate — 25 mg and 100 mg topiramate tablet 100 mg/day(50 mg bid) topiramate (maximum to 400 mg/day) Duration: maximum 52 weeks
  Arms: Topiramate

SUMMARY:
To assess the long-term effects of levetiracetam on retention rate in subjects with refractory partial onset seizure that are not fully controlled with 1 to 3 concomitant antiepileptic drugs, compared to topiramate as add-on therapy during 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects from 16 to 80 years, inclusive. Subjects under 20 years may only be included where legally permitted and ethically accepted
* Subjects with refractory epilepsy with partial onset seizure classifiable according to the International League Against Epilepsy (ILAE).
* Subjects having at least 2 partial onset seizures whether or not secondarily generalized during the 8 weeks historical baseline preceding V1 according to ILAE classification
* Subjects having at least 1 partial onset seizures whether or not secondarily generalized per 4 weeks preceding V2 according to ILAE classification
* Subjects with each interval of partial onset seizures less than 6 weeks during entire 12 weeks (8 weeks preceding V1 and 4 weeks preceding V2)
* Subjects being uncontrolled while treated by 1 to 3 permitted concomitant AEDs.
* Permitted concomitant AEDs having been stable and at optimal dosage for the subject from at least 4 week before V1 and during 4 weeks preceding V2 and expected to be kept stable during the Treatment Period.

Exclusion Criteria:

* Subjects presenting any generalized epilepsies classified as type II according to the ILAE classification (ref to publication from 1981)
* Subjects suffering from epilepsies and syndromes undetermined whether focal or generalized (classification III according to the ILAE classification)
* Subjects suffering from special syndromes (classification IV according to the ILAE classification)
* History or occurring only in clusters (too frequently or indistinctly separated to be reliably counted) before V2.
* Presence of exclusively type IA non-motor seizures.
* History or presence of status epilepticus within last 3 months preceding V1 or during Baseline
* History or presence of known pseudo-seizures
* Subjects who are currently on vigabatrin. (Subjects who received vigabatrin in the past and have a normal visual field test are allowed.)
* Subject taking 1 or more of the following medications on a regular basis within 28 days prior to Visit 1: antipsychotics drugs, and psychostimulant (amphetamine derivatives)

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2010-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — 1 877 822 9493 (UCB)
Locations (24):
- South Korea (24):
  - 14, Busan
  - 21, Busan
  - 8, Busan
  - 9, Busan
  - 12, Daegu
  - 13, Daegu
  - 10, Daejeon
  - 25, Daejeon
  - 15, Gwangju
  - 7, Incheon
  - 11, Kyunggi-Do
  - 19, Kyunggi-do
  - 23, Kyunggi-Do
  - 24, Kyunggi-Do
  - 16, Seoul
  - 17, Seoul
  - 18, Seoul
  - 1, Seoul
  - 2, Seoul
  - 3, Seoul
  - 4, Seoul
  - 5, Seoul
  - 6, Seoul
  - 22, Ulsan

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 447 subjects were screened, 343 subjects were randomized.
Pre-assignment Details: Participant Flow refers to the Randomized Set which consists of all subjects who were randomized in this study.
Period: Overall Study
Arm/Group | Levetiracetam | Topiramate
Started | 177 | 166
Completed | 111 | 100
Not Completed | 66 | 66
Not completed — Lack of Efficacy | 8 | 8
Not completed — Protocol Violation | 13 | 8
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 18 | 17
Not completed — Other Reason | 13 | 10
Not completed — SAE, non-fatal | 0 | 4
Not completed — AE, non-serious non-fatal | 13 | 17
Not completed — SAE, non-fatal+AE, non-serious non-fatal | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Characteristics refers to the Safety Set which consists of all subjects who were randomized and received at least 1 dose of trial medication.
Arm/Group | Levetiracetam | Topiramate | Total Title
Number analyzed (Participants) | 177 | 166 | 343
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 0 | 4
  Between 18 and 65 years | 165 | 162 | 327
  >=65 years | 8 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (13.6) | 39.7 (11.8) | 40.3 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 64 | 135
  Male | 106 | 102 | 208

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Continuing the Allocated Investigational Treatment From the First Study Treatment Intake to Week 52, After the Beginning of Investigational Treatment With Levetiracetam Compared to Topiramate
Time Frame: From Baseline to Week 52
Population: The Full Analysis Set (FAS) consisted of all subjects in the Safety Set who returned at least 1 post-baseline seizure diary.
Measure: Number; unit: percentage of subjects
Groups:
- Levetiracetam (Full Analysis Set): 250 mg and 500 mg levetiracetam tablet; titration from 1000 mg/day (500 mg bid) to 3000 mg/day (1500 mg bid) levetiracetam with treatment duration up to 52 weeks
- Topiramate (Full Analysis Set): 25 mg and 100 mg topiramate tablet; titration from 100 mg/day (50 mg bid) to 400 mg/day (200 mg bid) topiramate with treatment duration up to 52 weeks
Arm/Group | Levetiracetam (Full Analysis Set) | Topiramate (Full Analysis Set)
Number analyzed (Participants) | 176 | 166
percentage of subjects | 59.1 | 56.6
Statistical Analysis 1: Comparison: Levetiracetam (Full Analysis Set) vs Topiramate (Full Analysis Set); The Odds Ratio (OR) for LEV vs TPM is based on logistic regression modeling of subject retention by treatment and center pooling category. A profile likelihood confidence interval for the OR is presented; Test type: Superiority or Other; p = 0.7007, Regression, Logistic — P-value is from likelihood ratio test of treatment group regression coefficient against 0; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.7 to 1.7]

2. Secondary Outcome: Number of Subjects With at Least One Adverse Event Reported During the Trial Period From Baseline to Week 52
Time Frame: From Baseline to Week 52
Population: The Safety Set (SS) consists of all subjects who were randomized and received at least 1 (partial) dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Levetiracetam | Topiramate
Number analyzed (Participants) | 177 | 166
Participants | 125 | 128

3. Secondary Outcome: Time From the First Study Treatment Intake to Drug Discontinuation Due to Adverse Event (AE)
Time Frame: From Baseline to Week 52
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: month
Arm/Group | Levetiracetam | Topiramate
Number analyzed (Participants) | 177 | 166
month | NA [NA to NA] — For time to Study Drug Discontinuation due to AE, Kaplan-Meier estimation of event-free subjects does not fall to or below 75%, therefore no first quartile, median or third quartile of the time to event could be estimated in either group. | NA [NA to NA] — For time to Study Drug Discontinuation due to AE, Kaplan-Meier estimation of event-free subjects does not fall to or below 75%, therefore no first quartile, median or third quartile of the time to event could be estimated in either group.

4. Secondary Outcome: Median Percent Reduction in the Weekly Partial Onset Seizure (POS) Frequency From Baseline During the Total Treatment Period From Baseline to Week 52
Description: Reduction from baseline was defined as baseline value minus post-baseline value and therefore is the negative of the change from baseline value.
Time Frame: From Baseline to Week 52
Population: The Full Analysis Set (FAS) consists of all subjects in the Safety Set (SS) who returned at least 1 postbaseline seizure diary.
Measure: Median (Inter-Quartile Range); unit: percent reduction
Arm/Group | Levetiracetam (Full Analysis Set) | Topiramate (Full Analysis Set)
Number analyzed (Participants) | 174 | 165
percent reduction | 74.47 [38.00 to 96.28] | 67.86 [29.21 to 87.24]

5. Secondary Outcome: Responders Defined as Number of Subjects With at Least 50 % Reduction in the Weekly POS Frequency From Baseline During the Total Treatment Period From Baseline to Week 52
Time Frame: From Baseline to Week 52
Population: The Full Analysis Set (FAS) consists of all subjects in the SS who returned at least 1 postbaseline seizure diary.
Measure: Number; unit: responders
Arm/Group | Levetiracetam (Full Analysis Set) | Topiramate (Full Analysis Set)
Number analyzed (Participants) | 174 | 165
responders | 120 | 107

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from Visit 1 (Week -4) until final Visit 12 (Week 53).
Description: The Safety Set (SS) consisted of all subjects who were randomized and received at least 1 (partial) dose of study medication.
Arm/Group | Levetiracetam | Topiramate
Serious Adverse Events (participants affected / at risk) | 10/177 | 15/166
Other Adverse Events (participants affected / at risk) | 86/177 | 91/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (N=177) | Topiramate (N=166)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 5 (6)
Stupor (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (N=177) | Topiramate (N=166)
Dyspepsia (Gastrointestinal disorders) | 9 (10) | 7 (8)
Nausea (Gastrointestinal disorders) | 9 (11) | 10 (10)
Nasopharyngitis (Infections and infestations) | 24 (32) | 16 (22)
Weight decreased (Investigations) | 3 (3) | 17 (19)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 26 (32)
Somnolence (Nervous system disorders) | 36 (40) | 20 (21)
Dizziness (Nervous system disorders) | 30 (47) | 24 (29)
Headache (Nervous system disorders) | 17 (24) | 24 (25)
Tremor (Nervous system disorders) | 9 (9) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 9 (9)
Paraesthesia (Nervous system disorders) | 2 (2) | 16 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days